CLINICAL TRIAL: NCT00210366
Title: Salvage Therapy With Idarubicin in Immunocompetent Patients With Relapsed or Refractory Primary Central Nervous System Lymphomas
Brief Title: Salvage Therapy With Idarubicin in Relapsing CNS Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to slow accrual
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: International Extranodal Lymphoma Study Group, IELSG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG21
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Idarubicin

INTERVENTIONS:
Drug: Idarubicin

SUMMARY:
The main objective of the trial is to assess the therapeutic activity of idarubicin as salvage treatment in patients with recurrent or progressive lymphoma in the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-Hodgkin's lymphoma
* Disease exclusively localised into the CNS at first diagnosis and failure
* Progressive or recurrent disease
* Previous treatment with HDMTX containing CHT and/or RT
* Presence of at least one target lesion, bidimensionally measurable
* Age 18 - 75 years
* ECOG performance status < 3 (Appendix 1).
* No known HIV disease or immunodeficiency
* HBsAg-negative and Ab anti-HCV-negative patients.
* Adequate bone marrow function (plt > 100000 mm3, Hb > 9 g/dl, ANC > 2.000 mm3)
* Adequate renal function (serum creatinine < 2 times UNL)
* Adequate hepatic function (SGOT/SGPT < 3 times UNL, bilirubin and alkaline phosphatase < 2 times UNL)
* Adequate cardiac function (VEF ≥ 50%)
* Absence of any psycological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Non-pregnant and non-lactating status for female patients. Adequate contraceptive measures during study participation for sexually active patients of childbearing potential.
* No previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-site of the cervix and basal or squamous cell carcinoma of the skin and of other neoplasms without evidence of disease since at least 5 years.
* No concurrent treatment with other experimental drugs.
* Informed consent signed by the patient before registration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-11; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
objective response to treatment

SECONDARY OUTCOMES:
duration of response
overall survival
acute side effects of idarubicin

CONTACTS AND LOCATIONS:
Overall Officials: Andres JM Ferreri, MD, Study Chair — San Raffaele Hospital - HSR Servizio di radiochemioterapia
Locations (1):
- Servizio Radiochemioterapia - Ospedale San Raffaele, Milan, Milan, Italy

REFERENCES:
- See also: Click here for more information about this study — http://www.ielsg.org